CLINICAL TRIAL: NCT03799341
Title: Electrophysiological Predictors and Indicators of Contingency Management Treatment Response
Brief Title: Neurocognitive Factors in Substance Use Treatment Response: The Ways of Rewarding Abstinence Project
Acronym: WRAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NURA-002-18S; CX001807-01A1 (Other Grant/Funding Number: VA CSR&D)
Record Dates: First submitted 2019-01-07; First posted 2019-01-10 (Actual); Results first posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Cocaine Use Disorder
Keywords: Cocaine-Related Disorders; Contingency Management; Reward; Choice Behavior; Executive Function; Precision Medicine; Evidence-Based Practice; Prospective Thinking; Electroencephalography; Event-Related Potentials; Functional Connectivity
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to receive: (1) 12 weeks of TangiblePBCM (n = 70) or (2) 12 weeks of VoucherPBCM (n = 70). CM recipients will also be followed for 6 months post treatment. The proposed design enables evaluation of CM outcome predictors within 140 CM recipients - both with respect to initial treatment response and longer term (6 month) outcomes. All participants will receive a Baseline Assessment prior to the 12 Week Treatment interval, as well as a Follow-up Assessment at the conclusion of this period. Data from Baseline and Follow-up Assessments will enable longitudinal analysis of treatment-related change in EEG and cognitive-behavioral measures in treatment adherent versus treatment non-adherent subgroups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tangible Prize-Based Contingency Management (TangiblePBCM) (Experimental): For participants assigned to TangiblePBCM, prize draws resulting in one or more small, large, or jumbo wins will result in access to a prize cabinet stocked with small, medium, large, and jumbo financial incentive items. Medium incentive items are included for selection in the event that a patient draws several small prize slips on the same day and are considered equivalent to 4 small prizes. Selection of specific prize items will be informed by patient preference and items will be restocked at least every 2 weeks. The prize cabinet will be open during TangiblePBCM sessions such that prize items are readily visible. Selection of prizes, maintenance of the prize cabinet, and policies regarding prize redemption will follow published guidance on administration of TangiblePBCM within the context of research protocols.
  Interventions: Behavioral: Prize-Based Contingency Management; Behavioral: Treatment As Usual Outpatient Substance Use Treatment
- Voucher Prize-Based Contingency Management (VoucherPBCM) (Experimental): For participants assigned to VoucherPBCM, prize draws resulting in one or more small, large, or jumbo wins will be reinforced with VA Canteen vouchers in the specified incentive range (i.e., small, large, or jumbo).
  Interventions: Behavioral: Prize-Based Contingency Management; Behavioral: Treatment As Usual Outpatient Substance Use Treatment

INTERVENTIONS:
Behavioral: Prize-Based Contingency Management — Participants assigned to Prize-based Contingency
  Management (PBCM) conditions will receive PBCM as an adjunct to TAU. PBCM will involve twice weekly one-on-one sessions with a provider for 12-weeks. During each session, a urine specimen provided by the patient will be tested for cocaine using a point-of-care dip-test. Results of point-of-care testing will be shared with the patient and negative results will be reinforced with draws from a fish bowl containing 500 paper slips, 250 of which award small, large, or jumbo prizes (remaining slips deliver words of encouragement). Patients will be reinforced with a single prize draw for their first negative specimen; an additional prize draw will be added for each consecutive negative result (up to 8
  prize draws per session). Abstinence-contingent prize draws will be reset to one upon either a positive test result or unexcused, missed appointment.
Behavioral: Treatment As Usual Outpatient Substance Use Treatment — All participants will receive treatment as usual outpatient substance use services during the 12-week treatment interval. TAU will specifically entail recommended participation in at least two outpatient group and/or individual psychotherapy encounters per week within the Center for Treatment of Addictive Disorders (CTAD) at VA Pittsburgh Healthcare System. Participants will additionally continue any previously prescribed pharmacotherapy for substance use and/or other mental health conditions, if applicable.

SUMMARY:
The proposed work will investigate changes in brain signaling and cognitive functioning that support recovery from addiction, as well as use of pretreatment neurocognitive functioning to inform substance use treatment planning. Substance use disorders are prevalent amongst Veterans. Cocaine addiction, in particular, has been shown to complicate treatment of other high priority behavioral health problems in the Veteran population (e.g., PTSD, opioid addiction). While there are currently no approved medications to support recovery from cocaine addiction, research indicates that Contingency Management (CM) - a behavioral intervention for cocaine users - can be effective. However, individual responses are variable and long-term benefits are limited. This CDA will test a new model of how CM works by examining brain-based predictors and indicators of treatment response. Results will have immediate implications for measurement-based implementation of existing CM variants within the VA, supporting access to the version of CM that is best aligned with each Veteran's needs.

DETAILED DESCRIPTION:
Electrophysiological methods, including event-related potential and functional connectivity approaches, have potential to clarify mechanisms of substance use treatment response and characterize individual differences therein. Veterans are disproportionately affected by disorders of addiction, of which cocaine use disorder (CUD) is particularly problematic due to high relapse rates and the absence of approved pharmacotherapy options. Behavioral interventions for CUD have therefore become an important focus and Contingency Management (CM) has emerged as the best-supported approach. CM involves reinforcing cocaine abstinence (established through objective testing) with reliable, short-term reward, such as chances to win prizes (i.e., Prize-Based CM or PBCM). Given robust empirical support, nationwide dissemination of PBCM has been supported by a VHA initiative since 2011. However, PBCM response rates are variable and long-term benefits are limited - problems magnified by the cost of implementation with respect to staffing and prizes. Measurement-based approaches to PBCM implementation have promise to improve the effectiveness and efficiency of CM programming but have not yet been investigated within the VA or considered in relation to promising neuromarkers. Importantly, two versions of PBCM are already utilized at VA sites and may differentially benefit individuals with distinct neurocognitive profiles. Specifically, VA PBCM programs employ either abstract (voucher prize) or concrete (tangible prize) incentives, the latter of which may more effectively incentivize abstinence in Veterans with poor future-oriented thinking and planning ability. While selection between existing PBCM variants currently reflects practical considerations only, pretreatment neurocognitive functioning could meaningfully and realistically inform clinical decision-making in this regard.

This project aims to advance measurement-based implementation of CM by testing a novel neurocognitive model with immediate implications for the use of abstract versus concrete PBCM incentives within the VA. Specifically, the future-minded decision-making (FMDM) model posits that CM scaffolds future-oriented goal representation and self-control to support abstinence during in the moment use-related decision-making. For individuals with greater FMDM impairment, concrete, readily-accessible incentives may be more effective than abstract voucher-based rewards (which require future-oriented thinking and planning to acquire value). To test this model, neurocognitive substrates of FMDM will be examined as predictors of differential treatment response in voucher (VoucherPBCM) versus tangible prize (TangiblePBCM) versions of PBCM. Treatment-related change in neural and cognitive-behavioral correlates of FMDM will also be evaluated in PBCM-adherent versus non-adherent subgroups. Veterans with CUD will be allocated to VoucherPBCM or TangiblePBCM conditions and followed for a 12-week treatment interval. Pre- and post-treatment electroencephalography (EEG) and cognitive-behavioral assessments will be used to measure FMDM-related constructs (working memory, self-control, future-oriented decision-making, future reward representation) and related neuromarkers. These measures will be investigated as predictors of differential treatment response in VoucherPBCM versus TangiblePBCM, as well as maintenance of gains during a post-treatment follow-up period. Change in FMDM-related neural and cognitive measures over the course of treatment will also be evaluated for evidence of neuroadaptation (e.g., changes in functional connectivity) and enhancement of FMDM function through PBCM. Taken together, results of the current research project will represent a first step toward precision implementation of CM within the VA.

ELIGIBILITY:
Inclusion Criteria:

* Military Veterans
* DSM-5 Criteria for Cocaine Use Disorder (Mild, Moderate, or Severe)
* Cocaine Use Within Past 60 Days
* Stated Goal of Cocaine Abstinence or Reduced Cocaine Use
* Normal or Corrected-to-Normal Vision
* Average or Corrected Hearing

Exclusion Criteria:

* History of Severe Traumatic Brain Injury, Seizure Disorder, or other Neurological Illness
* Severe or Unstable Medical or Psychiatric Condition
* Pregnant or Lactating Women
* Moderate-to-Severe Neurocognitive Impairment per Medical Record, SLUMS < 21, or Mini MoCA < 11
* In Ongoing Residential Treatment or Imminently Expected to Enter Residential Treatment During the Study Interval at Time of Screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah E. Forster, PhD, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (1):
- VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
If possible, a de-identified, anonymized dataset will be created and shared. However, specific arrangements for sharing have not yet been made and options for data sharing (for example, the availability of data repositories for electroencephalographic data files), as well as VA policies regarding data sharing may change over the course of the study. A detailed plan for data sharing will be developed and approved upon completion of data collection.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place through the VA Pittsburgh Healthcare System and other local sites serving Veterans with Substance Use Disorders. Methods included mailings, provider referrals, public advertisements, event info tables, EHR screening, and announcements during therapy groups. Recruitment began in November 2019 but was paused due to COVID-19 from March 17, 2020, to January 15, 2021. It resumed thereafter and continued until enrollment ended on August 31, 2023.
Pre-assignment Details: Before randomization, participants completed a pre-screening interview. Those eligible were invited to enroll and proceed to full screening. Participants subsequently completed a baseline assessment visit that included biospecimen testing, interviews, questionnaires, cognitive-behavioral tasks, and an electroencephalography (EEG) session. Of the 122 unique Veterans prescreened, 63 met initial eligibility criteria and were enrolled in the study, with 45 subsequently proceeding to randomization.
Groups:
- Tangible Prize-Based Contingency Management (TangiblePBCM): Participants in this condition will receive Prize-Based Contingency Management (PBCM) as an adjunct to treatment as usual (TAU). During twice-weekly sessions, urine samples will be tested for cocaine, and each negative result earns the participant draws from a bowl of 500 paper slips, 250 of which award small, large, or jumbo prizes (the remaining slips deliver words of encouragement). Each consecutive negative adds an additional draw (up to 8), while a positive or missed test resets the draw count.
  For participants assigned to TangiblePBCM, prizes are awarded in the form of tangible items, which are chosen from a physical "prize cabinet." Participants may redeem their draws for small, medium, large, or jumbo prizes, with medium prizes valued at approximately 5 small prizes. The cabinet is visible during sessions and restocked regularly, and the selection of prizes is guided by patient preference. All participants continue to receive their usual outpatient treatment and medications alongside PBCM.
- Voucher Prize-Based Contingency Management (VoucherPBCM): Participants in this condition will receive Prize-Based Contingency Management (PBCM) as an adjunct to treatment as usual (TAU). During twice-weekly sessions, urine samples will be tested for cocaine, and each negative result earns the participant draws from a bowl of 500 paper slips, 250 of which award small, large, or jumbo prizes (the remaining slips deliver words of encouragement). Each consecutive negative adds an additional draw (up to 8), while a positive or missed test resets the draw count.
  For participants assigned to VoucherPBCM, prize draws resulting in small, large, or jumbo wins are rewarded with VA Canteen vouchers of corresponding value. These vouchers can be redeemed at Veterans Canteen Service vendors, including the hospital cafeteria and Patriot Store.
- Treatment As Usual (TAU): A treatment-as-usual (TAU) arm was originally included in the study design but was discontinued early in the trial due to evidence that its inclusion adversely affected participant accrual and retention among treatment-seeking individuals with cocaine use disorder. Participants randomized to TAU received standard care without the addition of prize-based contingency management (PBCM). Although they were still required to submit urine samples twice weekly for testing, they did not receive therapeutic incentives based on their urinalysis results.
Period: 12-Week Treatment Interval
Arm/Group | Tangible Prize-Based Contingency Management (TangiblePBCM) | Voucher Prize-Based Contingency Management (VoucherPBCM) | Treatment As Usual (TAU)
Started | 22 | 19 | 4
Completed | 22 | 19 | 2
Not Completed | 0 | 0 | 2
Not completed — Withdrawal by Investigator | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Period: Post-Tx Evaluation Session
Arm/Group | Tangible Prize-Based Contingency Management (TangiblePBCM) | Voucher Prize-Based Contingency Management (VoucherPBCM) | Treatment As Usual (TAU)
Started | 22 | 19 | 2
Completed (The Post-Tx Evaluation Session was considered completed if one or more follow-up assessments for this visit were completed.) | 17 | 13 | 2
Not Completed | 5 | 6 | 0
Not completed — Lost to Follow-up | 4 | 4 | 0
Not completed — Declined or Unavailable | 1 | 2 | 0
Period: 6-Month Post-Tx Follow-Up Period
Arm/Group | Tangible Prize-Based Contingency Management (TangiblePBCM) | Voucher Prize-Based Contingency Management (VoucherPBCM) | Treatment As Usual (TAU)
Started (Please note that participants were permitted to enter the 6-Month Post-Treatment Follow-Up Period regardless of whether they completed the Post-Treatment Evaluation Session. As a result, the number of participants entering this period was the same as the number who completed the treatment period. TAU participants completed the study at the time of the Post-Treatment Evaluation Session and were therefore excluded from this phase of the study.) | 22 | 19 | 0
Completed | 9 | 9 | 0
Not Completed | 13 | 10 | 0
Not completed — Lost to Follow-up | 12 | 10 | 0
Not completed — Withdrawal by Investigator | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tangible Prize-Based Contingency Management (TangiblePBCM) | Voucher Prize-Based Contingency Management (VoucherPBCM) | Treatment As Usual (TAU) | Total
Number analyzed (Participants) | 22 | 19 | 4 | 45
Age, Continuous [Mean (Standard Deviation); unit: age in years] | 61.9 (7.2) | 57.5 (7.9) | 61.5 (4.4) | 60.0 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 3
  Male | 20 | 18 | 4 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 21 | 18 | 4 | 43
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 18 | 12 | 4 | 34
  White | 3 | 7 | 0 | 10
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 22 | 19 | 4 | 45
% Self-Reported Pre-Treatment Cocaine-Abstinent Days [Mean (Standard Deviation); unit: % cocaine-abstinent days (past month)] — Values reflect retrospective reports of past-month substance use, obtained via the Timeline Follow-Back procedure at baseline. Notably, some participants were in controlled environments during this period, which may have led to inflated estimates of cocaine-abstinent days relative to what might be expected in the outpatient setting where PBCM was delivered in the current study.
  % cocaine-abstinent days (past month) | 84.0 (18.0) | 91.7 (10.9) | 83.7 (12.7) | 87.2 (15.1)
% Self-Reported Pre-Treatment Drug- and Alcohol-Abstinent Days [Mean (Standard Deviation); unit: % fully abstinent days (past month)] — Values reflect retrospective reports of past-month substance use, obtained via the Timeline Follow-Back procedure at baseline. Notably, some participants were in controlled environments during this period, which may have led to inflated estimates of drug and alcohol-abstinent days relative to what might be expected in the outpatient setting where PBCM was delivered in the current study.
  % fully abstinent days (past month) | 70.8 (30.2) | 71.2 (36.7) | 60.7 (41.7) | 70.1 (33.4)

OUTCOME MEASURES:

1. Primary Outcome: % Cocaine-Negative Urine Specimens Per Participant
Description: Percentage of cocaine-negative urine specimens during the 12-week treatment interval out of the total number possible, computed on a per-participant basis. The denominator was adjusted for participants for whom a full course of treatment could not be delivered due to suspension of face-to-face research activities during the COVID-19 pandemic. Denominators were similarly adjusted for 2 TAU participants who withdrew from the study during the 12-week treatment interval. Descriptive statistics represent the mean and standard deviation of the per-participant percentage of cocaine-negative urine specimens, computed across participants within each arm.
Time Frame: 12-Week Treatment Interval
Population: Results for the TAU arm are summarized using descriptive statistics but are omitted from statistical comparisons due to insufficient data (n = 4, with 2 out of 4 withdrawn from the study).
Measure: Mean (Standard Deviation); unit: % negative specimens per participant
Arm/Group | Tangible Prize-Based Contingency Management (TangiblePBCM) | Voucher Prize-Based Contingency Management (VoucherPBCM) | Treatment As Usual (TAU)
Number analyzed (Participants) | 22 | 19 | 4
% negative specimens per participant | 42.2 (37.4) | 59.1 (34.5) | 51.0 (18.8)
Statistical Analysis 1: Comparison: Tangible Prize-Based Contingency Management (TangiblePBCM) vs Voucher Prize-Based Contingency Management (VoucherPBCM); Test type: Other; p = 0.177, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Longest Duration of Cocaine Abstinence (LDCA)
Description: Longest period of objectively-verified abstinence from cocaine during treatment. It is noted that two TAU participants withdrew during the 12-week treatment interval. For these participants, the LDCA was computed for the pre-withdrawal period only.
Time Frame: 12-Week Treatment Interval
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: LDCA in days
Groups:
- Treatment As Usual: A treatment-as-usual (TAU) arm was originally included in the study design but was discontinued early in the trial due to evidence that its inclusion adversely affected participant accrual and retention among treatment-seeking individuals with cocaine use disorder. Participants randomized to TAU received standard care without the addition of prize-based contingency management (PBCM). Although they were still required to submit urine samples twice weekly for testing, they did not receive therapeutic incentives based on their urinalysis results.
Arm/Group | Tangible Prize-Based Contingency Management (TangiblePBCM) | Voucher Prize-Based Contingency Management (VoucherPBCM) | Treatment As Usual
Number analyzed (Participants) | 22 | 19 | 4
LDCA in days | 21.36 (27.87) | 34.95 (27.55) | 11.00 (19.34)
Statistical Analysis 1: Comparison: Tangible Prize-Based Contingency Management (TangiblePBCM) vs Voucher Prize-Based Contingency Management (VoucherPBCM); Test type: Other; p = 0.033, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: % Contingency Management (CM) Sessions Attended Per Participant (CM Groups Only)
Description: Percentage of CM treatment sessions attended out of the total number possible, computed on a per-participant basis. The denominator was adjusted for participants for whom a full course of treatment could not be delivered due to suspension of face-to-face research activities during the COVID-19 pandemic. Descriptive statistics represent the mean and standard deviation of the per-participant percentage of CM sessions attended, computed across participants within each arm.
Time Frame: 12-Week Treatment Interval
Measure: Mean (Standard Deviation); unit: % CM sessions attended per participant
Arm/Group | Tangible Prize-Based Contingency Management (TangiblePBCM) | Voucher Prize-Based Contingency Management (VoucherPBCM)
Number analyzed (Participants) | 22 | 19
% CM sessions attended per participant | 51.7 (33.2) | 68.0 (31.2)
Statistical Analysis 1: Comparison: Tangible Prize-Based Contingency Management (TangiblePBCM) vs Voucher Prize-Based Contingency Management (VoucherPBCM); Test type: Other; p = 0.126, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Total Non-CM Treatment Encounters Per Participant
Description: Number of non-CM, recovery-oriented treatment encounters during the 12-week treatment interval, computed on a per-participant basis. Encounters were documented in the electronic health record (VA encounters) and/or self-reported (non-VA encounters, including interactions with mutual support communities). Because this measure reflects the absolute number of non-CM treatment encounters per participant, only individuals with complete data for the 12-week period were included.
Time Frame: 12-Week Treatment Interval
Population: Only participants with complete data for the 12-week treatment period were included in this measure. Accordingly, two participants who withdrew early were excluded from the TAU arm, and one participant was excluded from the TangiblePBCM arm due to missing data. Results for the TAU arm are summarized using descriptive statistics but are omitted from statistical comparisons due to insufficient data (n = 4, with 2 out of 4 withdrawn from the study).
Measure: Mean (Standard Deviation); unit: count of encounters per participant
Arm/Group | Tangible Prize-Based Contingency Management (TangiblePBCM) | Voucher Prize-Based Contingency Management (VoucherPBCM) | Treatment As Usual (TAU)
Number analyzed (Participants) | 21 | 19 | 2
count of encounters per participant | 10.7 (15.8) | 12.5 (12.9) | 20.0 (24.0)
Statistical Analysis 1: Comparison: Tangible Prize-Based Contingency Management (TangiblePBCM) vs Voucher Prize-Based Contingency Management (VoucherPBCM); Test type: Other; p = 0.384, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: % Self-Reported Cocaine-Abstinent Days During Treatment
Description: Percentage of self-reported cocaine-abstinent days during the 12-week treatment interval, computed on a per-participant basis. Only participants with complete self-report data for the full treatment interval were included.
Time Frame: 12-Week Treatment Interval
Population: Two participants were excluded from each arm (TangiblePBCM, VoucherPBCM, TAU) due to missing self-reported substance use data (collected via timeline follow-back procedure) during the 12-week treatment interval. All participants included had complete self-report data for the full interval. Results for the TAU arm are summarized using descriptive statistics but are omitted from statistical comparisons due to insufficient data (n = 4, with 2 out of 4 withdrawn from the study).
Measure: Mean (Standard Deviation); unit: % cocaine abstinent days
Arm/Group | Tangible Prize-Based Contingency Management (TangiblePBCM) | Voucher Prize-Based Contingency Management (VoucherPBCM) | Treatment As Usual (TAU)
Number analyzed (Participants) | 20 | 17 | 2
% cocaine abstinent days | 86.0 (26.5) | 86.8 (24.4) | 81.7 (25.9)
Statistical Analysis 1: Comparison: Tangible Prize-Based Contingency Management (TangiblePBCM) vs Voucher Prize-Based Contingency Management (VoucherPBCM); Test type: Other; p = 0.308, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: % Self-Reported Drug- and Alcohol-Abstinent Days During Treatment
Description: Percentage of self-reported drug and alcohol-abstinent days during the 12-week treatment interval, computed on a per-participant basis. Only participants with complete self-report data for the full treatment interval were included.
Time Frame: 12-Week Treatment Interval
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: % drug and alcohol abstinent days
Arm/Group | Tangible Prize-Based Contingency Management (TangiblePBCM) | Voucher Prize-Based Contingency Management (VoucherPBCM) | Treatment As Usual (TAU)
Number analyzed (Participants) | 20 | 17 | 2
% drug and alcohol abstinent days | 72.6 (32.2) | 65.3 (39.6) | 56.4 (9.9)
Statistical Analysis 1: Comparison: Tangible Prize-Based Contingency Management (TangiblePBCM) vs Voucher Prize-Based Contingency Management (VoucherPBCM); Test type: Other; p = 0.976, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: % Self-Reported Stimulant-Abstinent Days at Post-Treatment (CM Groups Only)
Description: Percentage of self-reported stimulant-abstinent days during the 6 month post-treatment interval. For participants without complete data for the full 6-month post-treatment interval, the percentage of self-reported stimulant-abstinent days was computed based on the total number of days for which self-report data were available.
Time Frame: 6 Month Post-Treatment Interval
Measure: Mean (Standard Deviation); unit: % stimulant-abstinent days
Arm/Group | Tangible Prize-Based Contingency Management (TangiblePBCM) | Voucher Prize-Based Contingency Management (VoucherPBCM)
Number analyzed (Participants) | 19 | 15
% stimulant-abstinent days | 86.1 (27.8) | 92.1 (11.5)
Statistical Analysis 1: Comparison: Tangible Prize-Based Contingency Management (TangiblePBCM) vs Voucher Prize-Based Contingency Management (VoucherPBCM); Test type: Other; p = 0.920, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: % Self-Reported Drug- and Alcohol-Abstinent Days at Post-Treatment (CM Groups Only)
Description: Percentage of self-reported drug- and alcohol-abstinent days during the 6 month post-treatment interval. For participants without complete data for the full 6-month post-treatment interval, the percentage of self-reported stimulant-abstinent days was computed based on the total number of days for which self-report data were available.
Time Frame: 6 Month Post-Treatment Interval
Measure: Mean (Standard Deviation); unit: % drug and alcohol abstinent days
Arm/Group | Tangible Prize-Based Contingency Management (TangiblePBCM) | Voucher Prize-Based Contingency Management (VoucherPBCM)
Number analyzed (Participants) | 19 | 15
% drug and alcohol abstinent days | 70.9 (37.6) | 72.7 (34.4)
Statistical Analysis 1: Comparison: Tangible Prize-Based Contingency Management (TangiblePBCM) vs Voucher Prize-Based Contingency Management (VoucherPBCM); Test type: Other; p = 0.873, Wilcoxon (Mann-Whitney)

9. Other Pre Specified Outcome: Difference in Control-related Theta Synchronization From Baseline to Post-Treatment
Description: Theta synchronization between anterior cingulate cortex (Cz) and lateral prefrontal cortex (F3, F4, FC5, FC6) was measured to assess differences in functional connectivity between baseline and post-treatment (i.e., follow-up assessment conducted after the conclusion of the 12-week treatment interval) for high versus low conflict events. At each timepoint, phase locking value (PLV) was computed for 4 electrode pairs (Cz-F3, Cz-F4, Cz-FC5, Cz-FC6) across 3 stimulus conditions ranging from low to high conflict (Congruent, Intermediate-Incongruent, High-Incongruent) and for high-conflict error versus low-conflict correct responses in the Parametric Conflict Flankers task. A wavelet transformation isolated theta activity, and PLV was derived from normalized complex wavelet phases. PLV quantifies trial-to-trial phase synchrony (0-1), with 1 representing perfect synchrony. Descriptive data reported below represent the average PLV across the 4 electrode pairs.
Time Frame: Baseline and Post-Treatment Follow-up
Population: To accommodate the smaller final sample relative to the original target, analyses of neural and cognitive-behavioral outcomes were combined across arms. A revised analytic plan, approved prior to analysis, examined longitudinal differences by treatment engagement (attendance) and abstinence across arms.
Measure: Mean (Standard Deviation); unit: Phase Locking Value
Groups:
- All Participants With Pre/Post Data: All participants with data from both the baseline testing session and post-treatment testing session were included.
Arm/Group | All Participants With Pre/Post Data
Number analyzed (Participants) | 21
Phase Locking Value
  Baseline Congruent | 0.163 (0.096)
  Baseline Intermediate Incongruent | 0.173 (0.100)
  Baseline High Incongruent | 0.205 (0.098)
  Follow-Up Congruent | 0.158 (0.084)
  Follow-Up Intermediate Incongruent | 0.165 (0.083)
  Follow-Up High Incongruent | 0.200 (0.088)
  Baseline Correct | 0.169 (0.099)
  Baseline Error | 0.273 (0.146)
  Follow-Up Correct | 0.158 (0.086)
  Follow-Up Error | 0.245 (0.104)
Statistical Analysis 1: Comparison: All Participants With Pre/Post Data; Due to violations of normality assumptions, a non-parametric Aligned Rank Transform ANOVA was conducted, which does not permit inclusion of covariates. A median split approach was therefore used to examine the influence of Contingency Management session attendance. The design included 4 factors: time (2 levels), stimulus condition (3 levels), electrode pair (4 levels), and median split group membership (2 levels). Reported results reflect the interaction between time and median split group; Test type: Other; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: All Participants With Pre/Post Data; Due to violations of normality assumptions, a non-parametric Aligned Rank Transform ANOVA was conducted, which does not permit covariates. A median split approach was therefore used to examine the influence of self-reported cocaine abstinence during treatment. The design included 4 factors: time (2 levels), stimulus condition (3 levels), electrode pair (4 levels), and median split group membership (2 levels). Reported results reflect the interaction between time and median split group; Test type: Other; p < 0.001, ANOVA
Statistical Analysis 3: Comparison: All Participants With Pre/Post Data; Due to violations of normality assumptions, a non-parametric Aligned Rank Transform ANOVA was conducted, which does not permit inclusion of covariates. A median split approach was therefore used to examine the influence of Contingency Management session attendance. The design included 4 factors: time (2 levels), response accuracy (2 levels), electrode pair (4 levels), and median split group membership (2 levels). Reported results reflect the interaction between time and median split group; Test type: Other; p = 0.022, ANOVA
Statistical Analysis 4: Comparison: All Participants With Pre/Post Data; Due to violations of normality assumptions, a non-parametric Aligned Rank Transform ANOVA was conducted, which does not permit covariates. A median split approach was therefore used to examine the influence of self-reported cocaine abstinence during treatment. The design included 4 factors: time (2 levels), response accuracy (2 levels), electrode pair (4 levels), and median split group membership (2 levels). Reported results reflect the interaction between time and median split group; Test type: Other; p = 0.024, ANOVA

10. Other Pre Specified Outcome: Difference in Executive Working Memory From Baseline to Post-Treatment
Description: Difference in Brown-Peterson working memory scores between baseline and post-treatment (i.e., follow-up assessment conducted after the conclusion of the 12-week treatment interval). We will specifically use a modified Brown-Peterson test (Auditory Consonant Trigrams) for which both age- and Veteran-specific norms exist. Summary scores for this measure (including 9-, 18-, and 36-second delay conditions) can range from 0-45, with higher scores indicating improved executive working memory performance.
Time Frame: Baseline and Post-Treatment Follow-up
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: total score
Arm/Group | All Participants With Pre/Post Data
Number analyzed (Participants) | 27
total score
  Score at Baseline | 24.37 (7.82)
  Score at Follow-up | 24.78 (7.90)
Statistical Analysis 1: Comparison: All Participants With Pre/Post Data; No violations of normality assumptions were identified. A repeated measures ANOVA was conducted. To maintain consistency with other outcome measures, a median split approach was used to examine the potential influence of Contingency Management session attendance. The design included two factors: time (2 levels) and median split group membership (2 levels). Reported results reflect the interaction between time and median split group; Test type: Other; p = 0.973, ANOVA
Statistical Analysis 2: Comparison: All Participants With Pre/Post Data; No violations of normality assumptions were identified. A repeated measures ANOVA was conducted. To maintain consistency with other outcome measures, a median split approach was used to examine the potential influence of self-reported cocaine abstinence during the 12-week treatment interval. The design included two factors: time (2 levels) and median split group membership (2 levels). Reported results reflect the interaction between time and median split group; Test type: Other; p = 0.662, ANOVA

11. Other Pre Specified Outcome: Difference in Episodic Future Thinking Effect on Delay Discounting From Baseline to Post-Treatment
Description: Delay discounting was quantified using the hyperbolic discounting parameter (k), estimated separately for the Episodic Future Thinking (EFT) condition-with personally meaningful event tags anchoring delayed rewards-and the Standard condition without such tags. Values of k were natural log-transformed (ln(k)), with higher ln(k) indicating steeper discounting of delayed rewards, reflecting greater devaluation of future outcomes and a stronger preference for immediate gratification.
Time Frame: Baseline and Post-Treatment Follow-up
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ln(k) delay discounting parameter
Arm/Group | All Participants With Pre/Post Data
Number analyzed (Participants) | 28
ln(k) delay discounting parameter
  EFT ln(k) Baseline | -3.62 (2.15)
  Standard ln(k) Baseline | -2.42 (3.28)
  EFT ln(k) Follow-up | -3.36 (2.47)
  Standard ln(k) Follow-up | -2.77 (3.30)
Statistical Analysis 1: Comparison: All Participants With Pre/Post Data; Due to violations of normality assumptions, a non-parametric Aligned Rank Transform ANOVA was conducted, which does not permit inclusion of covariates. A median split approach was therefore used to examine the potential influence of Contingency Management session attendance. The design included 3 factors: time (2 levels), condition (2 levels), and median split group membership (2 levels). Reported results reflect the interaction between time, condition, and median split group; Test type: Other; p = 0.878, ANOVA
Statistical Analysis 2: Comparison: All Participants With Pre/Post Data; Due to violations of normality assumptions, a non-parametric Aligned Rank Transform ANOVA was conducted, which does not permit inclusion of covariates. A median split approach was therefore used to examine the potential influence of self-reported cocaine abstinence during treatment. The design included 3 factors: time (2 levels), condition (2 levels), and median split group membership (2 levels). Reported results reflect the interaction between time, condition, and median split group; Test type: Other; p = 0.645, ANOVA

ADVERSE EVENTS:
Time Frame: from enrollment until 6 months post-treatment, up to 12 months
Description: SAEs are relatively common among individuals with chronic cocaine use disorder, often due to cocaine's adverse effects on cardiovascular and mental health. SAEs occurring during the pre-randomization period are reported under the arm to which participants were ultimately assigned, when applicable. Participants could continue to randomization if still determined eligible. One participant hospitalized during pre-randomization was withdrawn prior to randomization and is therefore not included.
Arm/Group | Tangible Prize-Based Contingency Management (TangiblePBCM) | Voucher Prize-Based Contingency Management (VoucherPBCM) | Treatment As Usual (TAU)
All-Cause Mortality (participants affected / at risk) | 1/22 | 0/19 | 0/4
Serious Adverse Events (participants affected / at risk) | 5/22 | 5/19 | 1/4
Other Adverse Events (participants affected / at risk) | 0/22 | 0/19 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tangible Prize-Based Contingency Management (TangiblePBCM) (N=22) | Voucher Prize-Based Contingency Management (VoucherPBCM) (N=19) | Treatment As Usual (TAU) (N=4)
hospitalization due to cardiac symptoms (Cardiac disorders) | 1 (2) | 1 (1) | 1 (2) — Hospitalization for cardiac symptoms, which may occur in the context of cocaine use, other substance use, and/or an underlying medical condition. Not expected to be related to the study interventions, which are behavioral in nature.
hospitalization for psychiatric symptoms (Psychiatric disorders) | 3 (3) | 3 (5) | 0 (0) — Hospitalization due to exacerbation of psychiatric symptoms, which may occur in the context of cocaine use, other substance use, or an underlying psychiatric condition. Study interventions are not expected to increase the risk of such events.
initial or prolonged hospitalization due to stroke (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) — Initial or prolonged hospitalization resulting from stroke or other cerebrovascular event. Not expected to be related to study interventions, which are behavioral in nature.
hospitalization due to acute intoxication (General disorders) | 0 (0) | 2 (2) | 0 (0) — Hospitalization due to acute intoxication from cocaine or another substance, or for medically supervised detoxification following recent substance use. Study interventions supporting abstinence are not expected to increase the risk of such events.
hospitalization due to neurological symptoms (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Hospitalization for the treatment of new neurological symptoms and/or pre-existing conditions. Not expected to be related to study interventions, which are behavioral in nature.
hospitalization due to skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Hospitalization due to an acute skin infection. Not expected to be related to study interventions, which are behavioral in nature.
accidental overdose (General disorders) | 1 (1) | 0 (0) | 0 (0) — Accidental overdose in the context of cocaine or other substance use. As the study interventions are designed to promote abstinence, they are not anticipated to elevate the risk of such events.

LIMITATIONS AND CAVEATS:
Predictive analyses of differential treatment response in Tangible vs. Voucher PBCM, a key aim of the broader project, fall outside typical RCT reporting standards and will be reported separately.

Recruitment was significantly impacted by the COVID-19 pandemic, resulting in a smaller sample than originally planned and reduced power.

Outcomes related to delay discounting and theta phase synchronization may vary depending on specific analytic and preprocessing choices.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-06-02): https://cdn.clinicaltrials.gov/large-docs/41/NCT03799341/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT03799341/ICF_001.pdf